CLINICAL TRIAL: NCT07188922
Title: Effect of Transition From Mechanical Ventilation to Spontaneous Breathing on Intraocular Pressure: A Prospective Observational Study in ICU Patients
Brief Title: Effect of Transition From Mechanical Ventilation to Spontaneous Breathing on Intraocular Pressure in ICU (VENT-IOP)
Acronym: VENT-IOP
Status: Completed | Type: Observational
Sponsor: Sevim Şenol Karataş (Other)
Responsible Party: Sponsor-Investigator, Sevim Şenol Karataş, Specialist in Anesthesiology, Elazıg Fethi Sekin Sehir Hastanesi
Organization: Elazıg Fethi Sekin Sehir Hastanesi (Other)
Other Study IDs: EFSH-ANES-2025-09-VENT
Record Dates: First submitted 2025-09-16; First posted 2025-09-23 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Mechanical Ventilation
Keywords: Intraocular Pressure (IOP); Mechanical Ventilation; Spontaneous Breathing; Ventilator Weaning; Intensive Care Unit; Prospective Observational Study
MeSH Terms: interventions — Intraocular Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ICU Weaning Cohort: Adult patients in the intensive care unit undergoing transition from mechanical ventilation to spontaneous breathing. Intraocular pressure will be measured before and after the transition without any additional intervention beyond routine care.
  Interventions: Other: Non-invasive intraocular pressure measurement during ventilator weaning Description: Intraocular pressure will be measured using a portable non-invasive tonometer before and after the transition from

INTERVENTIONS:
Other: Non-invasive intraocular pressure measurement during ventilator weaning Description: Intraocular pressure will be measured using a portable non-invasive tonometer before and after the transition from — Intraocular pressure will be measured using a portable non-invasive tonometer before and after the transition from mechanical ventilation to spontaneous breathing. Measurements will be performed as part of routine clinical care and will not involve any experimental intervention.
  Other Names: Intraocular Pressure Measurement

SUMMARY:
This prospective, single-center observational study aims to evaluate the acute effects of transitioning from mechanical ventilation to spontaneous breathing on intraocular pressure (IOP) in intensive care unit patients. Forty adult patients receiving invasive mechanical ventilation and undergoing weaning will be enrolled. IOP will be measured non-invasively before and after the transition, without any intervention beyond routine clinical care. The primary objective is to determine whether spontaneous breathing after mechanical ventilation causes significant changes in IOP. Findings may provide insights into ocular physiology during weaning and contribute to the safe management of critically ill patients, particularly those with ocular risk factors.

DETAILED DESCRIPTION:
Mechanical ventilation is an essential life-supporting therapy for critically ill patients with respiratory failure. However, prolonged mechanical ventilation is associated with increased risks of complications, making the weaning process a critical step in intensive care management. During weaning, patients are transitioned from supported modes (such as SIMV or PSV) to spontaneous breathing modes (such as CPAP or T-tube). This transition leads to changes in thoracic pressure and venous return, which may in turn affect intracranial and intraocular pressures.

Intraocular pressure (IOP) is a key parameter for maintaining ocular perfusion and is influenced by systemic hemodynamics, respiratory patterns, and intrathoracic pressure changes. Previous studies have shown that posture, Valsalva maneuvers, and mechanical ventilation can alter IOP. However, evidence on the acute effects of transitioning from invasive mechanical ventilation to spontaneous breathing on IOP remains limited.

This prospective, observational, single-center study will be conducted in the intensive care unit of Elazığ Fethi Sekin City Hospital, Department of Anesthesiology and Reanimation. Forty adult patients receiving invasive mechanical ventilation and undergoing clinically indicated weaning will be enrolled. IOP will be measured non-invasively before and after the transition to spontaneous breathing, using portable tonometry, without the use of topical anesthesia. Measurements will be taken in both eyes, and average values will be recorded.

Demographic and clinical data, including age, sex, diagnosis, duration of ventilation, sedation status (RASS), and timing of mode transition, will also be collected. The primary endpoint is the difference in IOP before and after the transition. Statistical analysis will include paired t-test or Wilcoxon signed-rank test, depending on data distribution. Repeated measures ANOVA or Friedman test will be used when applicable, with significance set at p < 0.05.

This study does not involve any intervention or deviation from standard clinical care. All weaning procedures will be conducted according to routine ICU protocols. The findings of this study are expected to contribute to the understanding of ocular physiology during critical illness and may be particularly relevant for the safe management of patients with ocular comorbidities such as glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 85 years
* Admitted to intensive care unit (ICU) and receiving invasive mechanical ventilation
* Clinically scheduled for weaning and transition to spontaneous breathing
* Able to undergo intraocular pressure (IOP) measurement before and after transition
* Written informed consent obtained from the patient or legal representative

Exclusion Criteria:

* History of glaucoma, ocular hypertension, or previous eye surgery
* Active ocular infection or trauma
* Hemodynamic instability that prevents safe measurement
* Inability to obtain reliable IOP measurements
* Refusal of consent by patient or legal representative

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to the intensive care unit of Elazığ Fethi Sekin City Hospital, Department of Anesthesiology and Reanimation, who are receiving invasive mechanical ventilation and undergoing clinically indicated weaning.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2025-09-16 (Actual); Primary Completion 2025-10-16 (Actual); Study Completion 2025-10-16 (Actual)

PRIMARY OUTCOMES:
Change in Intraocular Pressure (IOP) Before and After Transition to Spontaneous Breathing | Within 2 hours before and within 2 hours after ventilator weaning (transition to spontaneous breathing)
  Intraocular pressure will be measured in both eyes using a portable non-invasive tonometer within 2 hours before and within 2 hours after the transition from mechanical ventilation to spontaneous breathing. The average value will be used for analysis. The primary endpoint is the difference in IOP values before and after the transition.

SECONDARY OUTCOMES:
Change in Mean Arterial Pressure (MAP) Before and After Transition to Spontaneous Breathing | Within 2 hours before and 2 hours after ventilator weaning
  Mean arterial pressure will be recorded within 2 hours before and within 2 hours after transition from mechanical ventilation to spontaneous breathing. Values will be compared to assess hemodynamic changes during weaning.
Change in Heart Rate Before and After Transition to Spontaneous Breathing | Within 2 hours before and 2 hours after ventilator weaning
  Heart rate will be monitored continuously. Measurements will be documented within 2 hours before and 2 hours after the transition to spontaneous breathing.

CONTACTS AND LOCATIONS:
Overall Officials: Sevim Şenol Karataş, Principal Investigator — Elazığ Fethi Sekin City Hospital, Department of Anesthesiology and Reanimation
Locations (1):
- Elazığ Fethi Sekin City Hospital, Elâzığ, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because this is a single-center observational study with a limited sample size. Only aggregate data will be analyzed and reported in publications. Sharing IPD is not planned in order to protect patient confidentiality and comply with local ethical regulations.

REFERENCES:
- [Background] Berdahl JP, Allingham RR, Johnson DH. Cerebrospinal fluid pressure is decreased in primary open-angle glaucoma. Ophthalmology. 2008 May;115(5):763-8. doi: 10.1016/j.ophtha.2008.01.013. PMID 18452762
- [Background] Esteban A, Anzueto A, Frutos F, Alia I, Brochard L, Stewart TE, Benito S, Epstein SK, Apezteguia C, Nightingale P, Arroliga AC, Tobin MJ; Mechanical Ventilation International Study Group. Characteristics and outcomes in adult patients receiving mechanical ventilation: a 28-day international study. JAMA. 2002 Jan 16;287(3):345-55. doi: 10.1001/jama.287.3.345. PMID 11790214
- [Background] Boles JM, Bion J, Connors A, Herridge M, Marsh B, Melot C, Pearl R, Silverman H, Stanchina M, Vieillard-Baron A, Welte T. Weaning from mechanical ventilation. Eur Respir J. 2007 May;29(5):1033-56. doi: 10.1183/09031936.00010206. PMID 17470624
- See also: Elazığ Fethi Sekin City Hospital, Department of Anesthesiology and Reanimation — https://elazigsehir.saglik.gov.tr/